CLINICAL TRIAL: NCT06031792
Title: A 2D and 3D Radiographic Assessment of the Healing Pattern Associated With Conventional and Piezoelectric Periradicular Endodontic Microsurgery
Brief Title: Radiographic Assessment of the Healing Pattern Associated With Periradicular Endodontic Microsurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KingAbdullahUH1
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Periapical; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: A randomized prospective clinical study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezo endodontic surgery (Experimental): Experimental: Piezo endodontic surgery The osteotomy will be applied under magnification with a surgical operating microscope (at the apical third of the root. Osteotomy will be done with the Piezosurgery touch
  Interventions: Procedure: Piezo endodontic surgery
- Conventional endodontic surgery (Experimental): Experimental: Conventional endodontic surgery The osteotomy will be applied under magnification with a surgical operating microscope at the apical third of the root. Osteotomy will be done with air motor high speed hand-piece and round bur with copious irrigation
  Interventions: Procedure: Conventional endodontic surgery

INTERVENTIONS:
Procedure: Piezo endodontic surgery — Osteotomy will be done with Piezosurgery touch. After the soft tissue curettage and uncovering the root apex, the last 3 mm of the root apex will be resected perpendicular to the long axis of the tooth using piezotome. apical preparation will be performed and Biodentine®retrograde filling material will be placed. The flap will be re-approximated and interrupted suture using non-absorbable monofilament suture will be applied. Finally, Post-operative parallel Digital view.
  Arms: Piezo endodontic surgery
Procedure: Conventional endodontic surgery — After the soft tissue curettage and exposure of the root apex, the osteotomy will be performed using a conventional surgical handpiece. The same steps will be followed to prepare and restore the root, as well as to reposition the flap.
  Arms: Conventional endodontic surgery

SUMMARY:
Endodontic periradicular microsurgery is a dental procedure to treat apical periodontitis in cases in which healing has not occurred after non-surgical treatment or if it is not feasible. Recent advances in techniques and materials have resulted in more predictable outcomes. Piezotome is a new and innovative device, but limited evidence is available regarding its use in endodontics. The aim of this study is to assess the healing pattern of conventional periradicular microsurgery and piezoelectric periradicular microsurgery in 2- Dimensional and 3-Dimensional imaging, and further to perform histological analysis for the presence, location, and arrangement of bacteria in the excised apical portion of the root canal system.

DETAILED DESCRIPTION:
After meeting the inclusion criteria, a total of 44 Patients in need of endodontic microsurgery with persistent symptoms after acceptable primary root canal treatment or failed retreatment with persistent symptoms/periapical lesions will be included in this study. Participants will be randomly allocated to group one; conventional periradicular surgery or group two; piezoelectric periradicular microsurgery. A preoperative digital periapical and limited view cone beam computed tomography (CBCT) radiographs will be taken for each patient. At 12-18 months recall visit a second digital periapical radiograph and limited view CBCT will be taken. All images will be evaluated on high-definition LCD display with installed ImageJ software and CBCT software, and window settings will be fixed for all cases. Radiographs will be evaluated by two calibrated dentists. The excised root tip with their surrounding tissues will be fixed immediately after harvesting for 24 hours at 4 °C by immersion in 1% glutaraldehyde and 1% formaldehyde and referred to histopathologic laboratory. Fixed specimens will be demineralized in 10% formic acid and processed. Serial sectioning with hematoxylin and eosin staining will be done to locate the areas with the most severe reactions. In addition, the Taylor modification of the Brown-Brenn staining will be used to detect the presence of bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit patients
* Age (18-65 )
* Teeth that are periodontally healthy
* Coronally sealed root canal treated teeth

Exclusion Criteria:

* Patients with an active systematic disease that may affect the short- and long-term outcomes or restrict surgical intervention
* Emotionally distressed patients
* Patients who had received analgesics or antibiotics prior to surgery will be postponed
* Cases where orthograde endodontic treatment is feasible, will be retreated at the post-graduate clinics and not included in this study
* Teeth with poor prognosis (e.g., non-restorable, vertical root fracture, short roots, non-strategic tooth, endo-perio lesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Healing | to measure periapical lesion through study completion, an average of 1 year
  To compare conventional and piezotome endodontic apical surgery in terms of healing using 2-Dimensional and 3-Dimensional imaging CBCT.
Histological outcome | one sample is taken and compared immediately after surgery
  To correlate histological findings with clinical observation and radiographic findings for failed root canal treated teeth presenting

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No